CLINICAL TRIAL: NCT03960294
Title: Evidence-Based e-Health Solutions for Youth With Mental Illness - Phase II
Brief Title: DOZE Sleep App for Youth With Sleep Disturbance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Colleen Carney, Associate Professor, Toronto Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 348431
Record Dates: First submitted 2019-05-05; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Insomnia
Keywords: Insomnia; Adolescents; Young Adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DOZE Users (Experimental): Adolescents and young adults (AYAs) using DOZE for sleep disturbance.
  Interventions: Other: DOZE Sleep App

INTERVENTIONS:
Other: DOZE Sleep App — DOZE is an evidence-based cognitive behavioural therapy for insomnia app created specifically for use with adolescents and young adults.

SUMMARY:
Insomnia is a highly prevalent problem among adolescents and young adults (AYAs) with mental health issues. Although evidence-based treatments to quickly address insomnia exist, access to such treatments is limited and there is very little research in AYAs. Furthermore, some of the sleep problems of AYA are unique (e.g., voluntary sleep restriction, circadian phase delay, very poor sleep hygiene), so pediatric and adult programs are not suitable for this age group. This study will test an innovative program that consists of an integrated smart phone application (app) and web self-management system ("DOZE") to help adolescents and young adults sleep better. The first phase of this project, now completed, involved interviewing primary stakeholders of the app (AYAs) to evaluate a low-fidelity prototype of the app and to gather information regarding their opinion about what tools participants would use to improve their health and/or sleep. Using the data from phase I, the investigators have created an app that is acceptable, useful and easy to use while meeting the needs of AYAs experiencing sleep problems. In this study, the investigators will conduct an open trial of the app with 145 AYAs to evaluate usability, acceptability, and sleep and corollary outcomes using a mixed methods design.

The investigators hypothesize:

1. That participants (AYAs) will find the app satisfactory and credible;
2. DOZE will effect sleep-related behaviour change;
3. DOZE will contribute to improvements in energy, mood, and perceived quality of life.

Exploratory analyses will also be conducted to evaluate which aspects of DOZE participants (AYAs) found most helpful.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 24 years
* Experiencing sleep disturbance

Exclusion Criteria:

* None

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Treatment Evaluation Questionnaire | Endpoint (week 4 or later)
  A quantitative questionnaire consisting of 5 questions evaluating treatment credibility. Scores range from 5 to 35, with higher scores indicating a more favourable evaluation of treatment.
Acceptability E-Scale | Endpoint (week 4 or later)
  A quantitative questionnaire, created for the purposes of this study, consisting of 6 questions assessing the acceptability of the app (helpfulness, usefulness, understandability, ease of use, enjoyment, and overall satisfaction) using a 5-point Likert scale. Scores range from 5 to 30, with higher scores indicating greater acceptability of the app.
Qualitative Assessment: Post-Test | Endpoint (week 4 or later)
  A qualitative questionnaire, created for the purposes of this study, consisting of 4 open-ended questions to obtain feedback on the app. Because of its qualitative nature, no scores are associated with this outcome; rather, this assessment will be used to receive open-ended feedback from the participants about the aspects of the app that they did and did not like.

SECONDARY OUTCOMES:
Google Analytics: time spent on each app page | Everyday for duration of study participation (i.e., week 0 to week 4 or later)
  Google Analytics will be used to track the time spent by each participant on each page/area of the app. This information will be used qualitatively to understand which aspects of the app were found least/most helpful.
Google Analytics: number of times app logged in | Everyday for duration of study participation (i.e., week 0 to week 4 or later)
  Google Analytics will be used to track the number of times each participant logged into the app. Greater adherence to app use (and daily sleep tracking) indicates greater acceptability of the app.
Google Analytics: number of times app used | Everyday for duration of study participation (i.e., week 0 to week 4 or later)
  Google Analytics will be used to track the number of times participants used the app. Greater app use indicates greater acceptability of the app. Google Analytics will provide a count of the number of times the app was accessed.
Google Analytics: number of quizzes completed | Everyday for duration of study participation (i.e., week 0 to week 4 or later)
  Google Analytics will be used to track the number of quizzes each participant completed. Quizzes are included in the app under the "Tips" heading, and include questions that related to chronotype, difficulty winding down, difficulty getting up, sleep drunkenness, trouble staying awake, and fatigue. Quizzes are an optional feature of the app which are used to provide participants with psychoeducation about these topics and how they relate to symptoms of sleep disturbance.
Sleep diary parameters | Everyday for duration of study participation (i.e., week 0 to week 4 or later)
  Data extracted from sleep diaries, including variability in bedtime, variability in rise time, total sleep time, total time in bed, sleep onset latency, wake after sleep onset, number of awakenings, naps
Center for Epidemiological Studies Depression Scale-Revised (9 items) | Baseline (week 0) and endpoint (week 4 or later)
  Scores range from 0 to 36, with higher scores indicating more severe depressive symptoms.
State-Trait Inventory of Cognitive and Somatic Anxiety | Baseline (week 0) and endpoint (week 4 or later)
  This measure includes two scales: a state scale (with scores ranging from 21 to 84) and a trait scale (with scores ranging from 21 to 84). Higher scores on both scales indicate more severe symptoms of anxiety.
Fatigue Severity Scale | Baseline (week 0) and endpoint (week 4 or later)
  A total score is computed by summing all of the items (range: 9 to 63) and dividing the score by the number of items to yield an item average. Average scores range from 1 to 7, with higher average scores indicating more impairment due to fatigue.
Cleveland Adolescent Sleepiness Scale | Baseline (week 0) and endpoint (week 4 or later)
  Scores range from 0 to 64, with higher scores indicating greater sleepiness.
Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) | Baseline (week 0) and endpoint (week 4 or later)
  Assesses health-related quality of life using 8 subscales: vitality, physical functioning, bodily pain, general, health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health. Items in which higher scores indicate better functioning are reverse scored when creating subscale scores. Subscale scores are converted to T scores ranging from 0 to 100, with higher scores indicating worse functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen E Carney, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gradisar M, Gardner G, Dohnt H. Recent worldwide sleep patterns and problems during adolescence: a review and meta-analysis of age, region, and sleep. Sleep Med. 2011 Feb;12(2):110-8. doi: 10.1016/j.sleep.2010.11.008. Epub 2011 Jan 22. PMID 21257344
- [Background] Sivertsen B, Harvey AG, Lundervold AJ, Hysing M. Sleep problems and depression in adolescence: results from a large population-based study of Norwegian adolescents aged 16-18 years. Eur Child Adolesc Psychiatry. 2014 Aug;23(8):681-9. doi: 10.1007/s00787-013-0502-y. Epub 2013 Nov 30. PMID 24292341
- [Background] Hicks RA, Fernandez C, Pellegrini RJ. Striking changes in the sleep satisfaction of university students over the last two decades. Percept Mot Skills. 2001 Dec;93(3):660. doi: 10.2466/pms.2001.93.3.660. PMID 11806582
- [Background] Yang CM, Wu CH, Hsieh MH, Liu MH, Lu FH. Coping with sleep disturbances among young adults: a survey of first-year college students in Taiwan. Behav Med. 2003 Fall;29(3):133-8. doi: 10.1080/08964280309596066. PMID 15206832
- [Background] Crowley SJ, Acebo C, Carskadon MA. Sleep, circadian rhythms, and delayed phase in adolescence. Sleep Med. 2007 Sep;8(6):602-12. doi: 10.1016/j.sleep.2006.12.002. Epub 2007 Mar 26. PMID 17383934
- [Background] Aoki H, Ozeki Y, Yamada N. Hypersensitivity of melatonin suppression in response to light in patients with delayed sleep phase syndrome. Chronobiol Int. 2001 Mar;18(2):263-71. doi: 10.1081/cbi-100103190. PMID 11379666
- [Background] Mindell JA, Kuhn B, Lewin DS, Meltzer LJ, Sadeh A; American Academy of Sleep Medicine. Behavioral treatment of bedtime problems and night wakings in infants and young children. Sleep. 2006 Oct;29(10):1263-76. PMID 17068979
- [Background] Owens JA, Rosen CL, Mindell JA. Medication use in the treatment of pediatric insomnia: results of a survey of community-based pediatricians. Pediatrics. 2003 May;111(5 Pt 1):e628-35. doi: 10.1542/peds.111.5.e628. PMID 12728122
- [Background] Stojanovski SD, Rasu RS, Balkrishnan R, Nahata MC. Trends in medication prescribing for pediatric sleep difficulties in US outpatient settings. Sleep. 2007 Aug;30(8):1013-7. doi: 10.1093/sleep/30.8.1013. PMID 17702271
- [Background] Boerner KE, Coulombe JA, Corkum P. Barriers and facilitators of evidence-based practice in pediatric behavioral sleep care: qualitative analysis of the perspectives of health professionals. Behav Sleep Med. 2015;13(1):36-51. doi: 10.1080/15402002.2013.838766. Epub 2013 Dec 23. PMID 24364693
- [Background] Clarke G, Harvey AG. The complex role of sleep in adolescent depression. Child Adolesc Psychiatr Clin N Am. 2012 Apr;21(2):385-400. doi: 10.1016/j.chc.2012.01.006. PMID 22537732
- [Background] Speth TA, Coulombe JA, Markovich AN, Chambers CT, Godbout R, Gruber R, Hall WA, Reid GJ, Stremler R, Weiss SK, Witmans M, Corkum PV. Barriers, facilitators, and usability of an Internet intervention for children aged 1 to 10 years with insomnia. Translational Issues in Psychological Science 1(1): 16-31, 2015.
- [Background] Espie CA, Kyle SD, Williams C, Ong JC, Douglas NJ, Hames P, Brown JS. A randomized, placebo-controlled trial of online cognitive behavioral therapy for chronic insomnia disorder delivered via an automated media-rich web application. Sleep. 2012 Jun 1;35(6):769-81. doi: 10.5665/sleep.1872. PMID 22654196
- [Derived] Carmona NE, Usyatynsky A, Kutana S, Corkum P, Henderson J, McShane K, Shapiro C, Sidani S, Stinson J, Carney CE. A Transdiagnostic Self-management Web-Based App for Sleep Disturbance in Adolescents and Young Adults: Feasibility and Acceptability Study. JMIR Form Res. 2021 Nov 1;5(11):e25392. doi: 10.2196/25392. PMID 34723820